CLINICAL TRIAL: NCT02670928
Title: Interventional Study of Active Weight Management in Patients With Type 2 Diabetes and Obesity in Routine Clinical Practice During 12 Months.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLAF237ARU05
Record Dates: First submitted 2016-01-13; First posted 2016-02-02 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Diabetes; lifestyle change; weight management; control of glycemic in HbA1C and FPG
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active group of patients (Active Comparator): Active group of patients underwent program of active lifestyle management (healthy nutrition, physical exercises, psychological counselling and classes on diabetes) in first 12 weeks of the study.
  Interventions: Behavioral: Lifestyle intervention
- Control group of patients (Experimental): Control group pf patients were being monitored for the same criteria as active group but did not take part in the lifestyle change management program.
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — Patients of active group were assigned to receive activities of the program for life style changes. Patients in control group were managed in frames of routine clinical practice. No any investigational drug therapy was used.

SUMMARY:
This study was aimed to achieve of long-term weight loss in T2DM patients by use of comprehensive lifestyle changes program, providing patients with structured diet, exercise plan, group behavioral support and group education. Additionally the study was designed to establish reduction of the body weight leads to the improvement of glycemic and lipid metabolism, and also reducing blood pressure level. The study was also directed to show that lifestyle changes program in T2DM patients can lead to decreasing of hospitalization rate and healthcare consumption. In order to demonstrate a change from standard of care, data were to be collected from a parallel cohort from the same centers.

DETAILED DESCRIPTION:
Patients of active group were assigned to receive activities of the program for life style changes. Patients in control group were managed in frames of routine clinical practice. No any investigational drug therapy was used.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent. Written informed consent must be obtained before any assessment is performed.

  •≥ 18 years
* Type 2 diabetes
* The Body Mass Index is from 28 to 40 kg/m^2

Exclusion Criteria:

* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation.
* Type 1 diabetes
* Proliferative retinopathy
* Renal impairment: serum creatinine >1.5 mg/dL, creatinine clearance < 40 ml/min and/or proteinuria
* The lack of ability to perform the physical exercises due to the orthopedic or cardiovascular disorders
* Chronic alcoholism, acute alcoholic intoxication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Russia (2):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the following jurisdiction: Russia (2 centers).
Period: Overall Study
Arm/Group | Active Group of Patients | Control Group of Patients
Started (All enrolled patients (Full Analysis Set and Safety Population)) | 100 | 30
Completed | 90 | 29
Not Completed | 10 | 1
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Miss 3 classes in a row in first 12 wks | 2 | 0

BASELINE CHARACTERISTICS:
Population: All patients in the active and control groups were included in the population of all enrolled patients, the safety population and the full analysis set (FAS).
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Group of Patients | Control Group of Patients | Total
Number analyzed (Participants) | 100 | 30 | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (10.2) | 60.6 (8.9) | 56.0 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 19 | 88
  Male | 31 | 11 | 42
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 99 | 29 | 128
  Oriental | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinically Significant Weight Reduction (>5%) Compared to Baseline at Month 12
Description: Number (portion) of patients in the active group and control group in whom the body weight decreased by at least 5% compared to Baseline values at 12 months of follow-up
Time Frame: Baseline, Month 12
Population: Full Analysis Set (FAS) using the Last Observation Carried Forward (LOCF) approach for imputing missing data. Only descriptive analysis done.
Measure: Number; unit: Participants
Arm/Group | Active Group of Patients | Control Group of Patients
Number analyzed (Participants) | 100 | 30
Participants
  Week 48 (Month 12) - Yes | 50 | 4
  Week 48 (Month 12) - No | 50 | 26

2. Secondary Outcome: Percentage of Patients Who Achieved a Decrease in Blood Pressure Values From Baseline at Month 12
Description: Decrease in blood pressure value was defined as at least 5 millimeters mercury (mmHg) in systolic and diastolic values in comparison to Baseline
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Active Group of Patients | Control Group of Patients
Number analyzed (Participants) | 100 | 30
Percentage of Participants | 55 | 40

3. Secondary Outcome: Percentage of Patients With Clinically Significant Weight Reduction (>5%) Compared to Baseline
Description: Number (portion) of patients achieved weight loss by at least 5% in comparison with Baseline at 3, 6, 9 months of follow-up
Time Frame: Baseline, Month 3, Month 6, Month 9, Month 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Active Group of Patients | Control Group of Patients
Number analyzed (Participants) | 100 | 30
Percentage of Participants
  Week 12 (Month 3) - Yes | 40 | 13.3
  Week 12 (Month 3) - No | 60 | 86.7
  Week 24 (Month 6) - Yes | 34 | 26.7
  Week 24 (Month 6) - No | 66 | 73.3
  Week 36 (Month 9) - Yes | 39 | 16.7
  Week 36 (Month 9) - No | 61 | 83.3
  Week 48 (Month 12) - Yes | 50 | 13.3
  Week 48 (Month 12) - No | 50 | 86.7

4. Secondary Outcome: Percentage Change From Baseline in Cholesterol at Month 12
Description: Analysis of percentage changes in lipid profile (cholesterol, mmol/l) compared to Baseline at 12 months of follow-up
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Active Group of Patients | Control Group of Patients
Number analyzed (Participants) | 100 | 30
Percent change | -9.44 (2.792) | -8.00 (3.339)

5. Secondary Outcome: Percentage Change From Baseline in Triglycerides at Month 12
Description: Analysis of percentage in lipid profile (triglycerides, mmol/l) compared to Baseline at 12 months of follow-up
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Active Group of Patients | Control Group of Patients
Number analyzed (Participants) | 100 | 30
Percent change | -0.479 (0.1136) | 0.481 (0.2468)

6. Secondary Outcome: Percentage Change From Baseline in Lipid Protein of High and Low Density at Month 12
Description: Analysis of percentage in lipid profile (LDL, mmol/l and HDL, mmol/l) compared to Baseline at 12 months of follow-up
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Active Group of Patients | Control Group of Patients
Number analyzed (Participants) | 100 | 30
Percent change
  Low Density Lipoprotein (LDL) | -6.76 (4.649) | -11.54 (4.641)
  High Density Lipoprotein (HDL) | 17.46 (10.967) | 12.68 (6.089)

7. Secondary Outcome: Percentage of Participants With Change From Baseline in Quality of Life (QoL) at Month 12
Description: Patients were asked 'When did blood sugar level decrease most recently?' and the responses were reported on a Change in Quality of Life (QoL) expressed in percents using the Novartis survey in hypoglycemia and scale of individual perception of PhA (Scale of Borg)
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Active Group of Patients | Control Group of Patients
Number analyzed (Participants) | 90 | 29
Percentage of participants
  During last week | 5.6 | 3.4
  From 1 week to 1 month ago | 1.1 | 3.4
  From 1 to 6 month ago | 16.7 | 17.2
  More than 6 months ago and within last 12 months | 11.1 | 6.9
  More than 12 months ago | 11.1 | 6.9
  No episode of blood sugar level decrease | 54.4 | 62.1

8. Secondary Outcome: Percentage Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Month 12
Description: Analysis of percentage changes in Glycosylated hemoglobin (HbA1c, %) levels compared to Baseline at 12 months follow-up
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Active Group of Patients | Control Group of Patients
Number analyzed (Participants) | 92 | 30
Percent change | 6.640 (1.152) | 7.687 (1.558)

9. Secondary Outcome: Percentage Change From Baseline in Fasting Plasma Glucose (FPG) at Month 12
Description: Analysis of percentage changes in Fasting Plasma Glucose (FPG, mmol/l) levels compared to Baseline at 12 months of follow-up
Time Frame: Basline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Active Group of Patients | Control Group of Patients
Number analyzed (Participants) | 100 | 30
Percent change | 1.55 (7.217) | -3.03 (5.079)

10. Secondary Outcome: Percentage Hange From Baseline in Body Mass Index (BMI) at Month 12
Description: Changes of Baseline in Body Mass Index (BMI) levels expressed in percents compared to Baseline at 12 months of follow-up
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Active Group of Patients | Control Group of Patients
Number analyzed (Participants) | 100 | 30
Percent change | 32.417 (3.940) | 33.190 (4.075)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). Each patient was assessed for up to 12 months.
Description: The Safety Set consisted of all patients in the active group who started participating in the lifestyle correction program and all patients in the control group for whom the observation was started
Arm/Group | Active Group of Patients | Control Group of Patients
All-Cause Mortality (participants affected / at risk) | 0/100 | 1/30
Serious Adverse Events (participants affected / at risk) | 6/100 | 2/30
Other Adverse Events (participants affected / at risk) | 0/100 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Active Group of Patients (N=100) | Control Group of Patients (N=30)
Acute Myiocardial Infarction (Cardiac disorders) | 1/1 (1) | 1/1 (1)
Myocardial Ischemia (Cardiac disorders) | 1/1 (1) | 0/0 (0)
Duodenal ulcer Haemorrhage (Gastrointestinal disorders) | 1/1 (1) | 0/0 (0)
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0/0 (0) | 1/1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 1/1 (1) | 0/0 (0)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1 (1) | 0/0 (0)
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1 (1) | 0/0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2015-07-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT02670928/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT02670928/SAP_001.pdf